CLINICAL TRIAL: NCT04325048
Title: Single-Arm Observational Study Designed to Clinically Evaluate Cordio Application in Adult Patients Positive to COVID-19
Brief Title: Clinical Evaluation of Cordio Application in Adult COVID-19 Virus Positive Patients
Status: Completed | Type: Observational
Sponsor: Cordio Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: COV001
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Coronavirus Infection
Keywords: COVID-19 positive
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cordio App — Adult patients positive to COVID-19 virus will record several predefined sentences via a smartphone / tablet and will answer questions via the app

SUMMARY:
Study on adult patients positive to COVID-19 virus. After signing informed consent and undergoing screening assessments, eligible patients will record few times a day several pre-defined sentences to the Cordio App installed in a smartphone/tablet.

The app will upload the vocal data to the sponsor's servers for analysis. The patient will record at hospital admittance (COVID-19 positive) until patient defined as COVID-19 negative and free of relevant clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years old
2. Diagnosed with COVID-19 positive patients according to medical center guidelines, with symptoms of cough and or dyspnea. Patients that diagnosed with pneumonia, should be confirmed by X-ray and/or CT.
3. Able to understand and provide written informed consent (manually or electronically or giving their consent via the telephone to the study investigator in case of isolated patients).

Exclusion Criteria:

1. Subjects, in the Investigator's opinion, unable to comply with the daily use of the application including mental disorders (e.g., depression, dementia).
2. Patients with severe alcohol or drug use.
3. Women who are pregnant or lactating.
4. Participating in another investigation therapy that may interfere with study results (according to investigator discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients, from medical center departments, ER, home/hotels hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Voice anaysis | 1-2 years
  patient voice that is recorded during the study will be anylaysis with specific algorithms

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Azzam, Prof, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No